CLINICAL TRIAL: NCT05193396
Title: A Multi-centre, Randomised, Double-blinded, Placebo Controlled 16-weeks Study to Compare the Effect of Hydrocortisone and Placebo in Patients With Giant Cell Arteritis (GCA)/ Polymyalgia Rheumatica (PMR) With Patient-reported Symptoms of Adrenal Insufficiency After Cessation of Glucocorticoid Treatment.
Brief Title: Hydrocortisone and Placebo in Patients With Symptoms of Adrenal Insufficiency After Cessation of Glucocorticoid Treatment
Acronym: REPLACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marianne Andersen (Other)
Collaborators: Aarhus University Hospital (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor-Investigator, Marianne Andersen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REPLACE; 2024-513822-53-00 (EU CTIS Number); 2020-006121-65 (EudraCT Number); journal no. 21/27119 (Other: Danish Data Protection Agency); project-ID: S-20210076 (Other: Regional Committees on Health Research Ethics for Southern Denmark)
Record Dates: First submitted 2022-01-02; First posted 2022-01-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-03

CONDITIONS: Adrenal Insufficiency; Polymyalgia Rheumatica (PMR); Giant Cell Arteritis (GCA)
Keywords: tertiary adrenal insufficiency
MeSH Terms: conditions — Adrenal Insufficiency; Polymyalgia Rheumatica; Giant Cell Arteritis | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blinded randomised placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and all study personnel are blinded for study medication (hydrocortisone or placebo)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RCT group - Placebo (Placebo Comparator): Included patients with an AddiQoL-30 score < 85 and/or short Synacthen test stimulated plasma cortisol levels > 100 and < 420 nmol/L that are radomized to recieve placebo tablets.
  Interventions: Drug: Placebo
- RCT group - Hydrocortisone (Active Comparator): Included patients with an AddiQoL-30 score < 85 and/or short Synacthen test stimulated plasma cortisol levels > 100 and < 420 nmol/L that are radomized to recieve hydrocortisone tablets.
  Interventions: Drug: Hydrocortisone
- Comparator group 1 (No Intervention): Patients with an AddiQoL-30 score > 85 and short Synacthen test stimulated plasma cortisol level > 420 nmol/L. Patients undergo baseline examination only.
- Comparator group 2 (No Intervention): Patients with pronounced adrenal insufficiency (short Synacthen test stimulated plasma cortisol levels < 100 nmol/L) - regardless of AddiQoL-30 score. These patients undergo baseline examination and commence open hydrocortisone replacement according to standard clinical practice.

INTERVENTIONS:
Drug: Hydrocortisone — Patients are randomized to oral hydrocortisone (10 mg twice daily) or placebo for 16 weeks.
  Arms: RCT group - Hydrocortisone
Drug: Placebo — Patients are randomized to oral hydrocortisone (10 mg twice daily) or placebo for 16 weeks.
  Arms: RCT group - Placebo

SUMMARY:
Cortisol, a glucocorticoid (GC) hormone secreted from the adrenal glands, is essential for survival. Cortisol also possesses anti-inflammatory actions and GC formulations (prednisolone) are used to treat many inflammatory diseases and conditions. Indeed, three percent of the Danish population (≈ 180.000 individuals) redeems at least one prescription of synthetic GC per year and at least 20,000 patients annually discontinue GC treatment. Pharmacological GC therapy suppresses endogenous cortisol production and thereby induce relative adrenal insufficiency (GIA). The risk of GIA as determined by the adrenal corticotrophic hormone (ACTH) stimulation test has previously been reported to ≈ 25 %, but testing after GC treatment is not routinely performed. Indeed, new evidence suggest that the risk of GIA after planned cessation of prednisolone treatment for polymyalgia rheumatic (PMR) or giant cell arteritis (GCA) is substantially lower, probably 2%. The reason for this discrepancy is undoubtedly selection bias in the previous publications and the use of inaccurate cortisol assays. At the same time, however, it was observed that 25% exhibited pronounced symptoms of adrenal insufficiency based on a questionnaire specific for detecting symptoms of adrenal insufficiency, the so-called AddiQoL-30. Concomitantly, the basal cortisol levels in the same group were significantly lower as compared to the group, who exhibited milder or no symptoms attributable to adrenal insufficiency. This observation aligns with the clinical experience that PMR/GCA patients often complain of fatigue after planned cessation of prednisolone treatment. This often occurs in the absence of objective symptoms or signs of residual PMR/GCA disease activity. The scenario has been designated as "the steroid withdrawal syndrome". This may represent a state of relative adrenal insufficiency prompted by long term, high dose prednisolone treatment. The proper way to tackle this clinical conundrum is to perform a proper randomized trial, which so far has not been conducted.

Therefore, investigators of this study will perform the first placebo-controlled randomised controlled trial (RCT) in patients with PMR and GCA after planned cessation of GC treatment. Investigators argue that neither watchful waiting nor routine hydrocortisone replacement are infallible. The study will be the first evidence-based guidance and aid to GIA patients and thus meet an important need for many thousand patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* A diagnosis of PMR or GCA in GC free remission for >2 week and <12 weeks after treatment with prednisolone (any dosage) for ≥12 weeks

Exclusion Criteria:

* Known primary or secondary adrenal insufficiency
* Known Cushing´s syndrome
* Heart failure (New York Heart Association class IV)
* Kidney failure with an estimated glomerular filtration rate <30 mL/min
* Liver cirrhosis
* Active cancer
* Known severe immune deficiency
* A history of psychiatric disease requiring treatment by a psychiatric department (for affective disorders only if within the last year before study entry)
* Alcohol consumption >21 units per week
* Planned major surgery during the study period at study entry
* Use of drugs that interfere with cortisol metabolism/measurements:
* Systemic oestrogen treatment within 1 month before study inclusion
* Strong CYP3A4 inhibitors or inducers
* Use of other glucocorticoid formulations: inhaled, intra-articular or intramuscular injections, creams European steroid group IV applied in genital area
* Permitted glucocorticoid formulations: eye-drops, nasal spray, creams European group I-III, and European group IV applied in non-genital area
* Inability to provide written informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Adrenal insufficiency symptoms | Screening and 16 weeks
  Symptoms measured by the Addison's disease-specific quality of life questionnaire (AddiQoL-30), which consists of 30 questions focusing on common symptoms of adrenal insufficiency related to quality of life. Each item belongs to one of following subthemes: fatigue, symptoms, emotions and miscellaneous. Each question can be scored from 1 (none of the time/strongly disagree) to 6 (all of the time/strongly agree) and yields a score between 1 - 4 arbitrary units. This adds up to a total score ranging from 30 (worst quality of life) to 120 (best quality of life).

SECONDARY OUTCOMES:
Patient-reported symptoms via mobile phone app - PRO-CTCAETM | Patients are asked daily throughout the study period.
  Symptoms of fatigue, nausea, dizziness, and "feeling generally unwell" assessed by the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAETM). Each symptom is evaluated in terms of frequency and severity with a score from 1 (never/nothing) to 5 (almost constant/very strong).
Patient-reported symptoms via mobile phone app - EMA-MFI | In situations of stress, participants are asked to answer the EMA items 5 times daily at semi-randomised time points, for 3 days.
  Four statements regarding diurnal fatigue based on the validated General Fatigue Scale from the Multidimensional Fatigue Inventory (MFI-20) adapted for Ecological Momentary Assessments (EMA). Each statement is answered by a visuel scale from left (yes, that is correct) to right (no, that is not correct).
Cushing quality of life (CushingQoL) | Baseline and 16 weeks
  Cushing quality of life (CushingQoL) is a disease-specific questionnaire for patients with endogenous cortisol excess. It consists of 12 items about mental and physical adverse effects of cortisol excess. The total score os normalised to a scale ranging from 0 (lowest quality of lige) to 100 (highest quality of life).
The short form 36 (SF-36) | Baseline and 16 weeks
  SF-36 is a genereic qeustionnaire evaluating general health perception with 36 items related to 8 dimensions: physical functioning for the limitation in performing all physical activities; role physical for problems with work or other daily activities; bodily pain; general health; vitality; social functioning; role emotional; and mental health.
Sleep Quality Scale (SQS) | Baseline and 16 weeks
  SQS is a single item questionnaire consisting of a numerical rating scale to evaluate the overall sleep quality over the last 7 nights. The scale is ranging from 0 (terrible sleep) to 10 (excellent sleep).
International Physical Activity Questionnaire, short form, 7 days (IPAQ-7s) | Baseline and 16 weeks
  The IPAQ-7s records types and intensity of physical activity. The questionnaire consists of seven open items covering 4 types of activity (energetic activity, moderate activity, walk, and sitting). The first three is measured in "number of days per week", "hours per day", and "minutes per day". The last activity (sitting) is measured in "hours per day" and "minutes per day".
Incidence of adrenal crises | 16 weeks
  Incidence of adrenal crises, including information on hospitalizations, number of sick days, diagnoses and therapy.
Cardiovascular health - Blood pressure | Baseline and 16 weeks
  Office blood pressure (OBP) and automated blood pressure (AOBP). Blood pressure measurements will be performed with (OBP) and without (AOBP) the presence of investigator. Unit is mmHg.
Cardiovascular health - PWV | Baseline and 16 weeks
  Arterial stiffness and pulse wave velocity (PWV). PVW is measured three times, unit is m/s.
Body composition - DXA scan | Only performed at baseline visit
  Body composition by dual X-ray absorptiometry (DXA) scan. Body composition is measured in the distribution of fat and lean mass in grams (g).
Bone quality - DXA scan | Only performed at baseline visit
  Bone quality by dual X-ray absorptiometry (DXA) scan. Bone mineral density (g/cm^2) and T-score of the lumbal spine and hip.
HR-pQCT | Only performed at baseline visit
  High-resolution peripheral quantitative computed tomography (HR-pQCT) in order to obtain three-dimensional BMD.
Muscle function and physical activity - Handgrip strength. | Baseline and 16 weeks.
  Handgrip strength is measured in kg using a hydraulic hand dynamometer.
Muscle function and physical activity - TUG | Baseline and 16 weeks.
  Timed Up and Go (TUG) test measures the time taken to stand up, walk three meters in a straight line, and immediately return to the chair.
Muscle function and physical activity - SPPB | Baseline and 16 weeks.
  The Short Physical Performance Battery including Chair Rising Test (SPPB) evaluates the lower extremity function of the patient.
Muscle function and physical activity - Actigraph | Baseline and 16 weeks, duration: 7 days
  Patients are asked to wear an accelerometer device on their non-dominant wrist to measure physical activity and sleep. Time of physical activity and sleep will be measured in minutes.
Muscle function and physical activity - Muscle power | Baseline and 16 weeks.
  The muscle power of the dominant arm and upper back, as well as elbow, hip, and knee extension and flexion, are evaluated by use of a exercise machine. Power is measured in watt.
Muscle function and physical activity - Isometric muscle strength | Baseline and 16 weeks.
  The isometric muscle strength of the dominant arm and upper back, as well as elbow, hip, and knee extension and flexion, are evaluated by use of a exercise machine. Strength is measured in kg.
Normalization of adrenal function evaluated by SST | Screening/Baseline and 16 weeks
  Short Synacthen® test. Cortisol is measured in nmol/L before (0 min) and after (30 min) administration of 1 ml Synacthen (0.25 mg/ml).

OTHER OUTCOMES:
Blood samples (unit: 10E12/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  Erythrocytes.
Blood samples (unit: fmol) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  MCH.
Blood samples (unit: 10E9/L). | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  Leokocytes; neutrophils; lymphocytes; monocytes; basophilocytes; eosinophils; metamyelocytes; thrombocytes.
Blood samples (unit: mmol/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  Hemoglobin; MCHC; glucose; glucose derived from HbA1c, cholesterol; HDL; LDL; non-HDL; triglycerid; calcium ion, free.
Blood samples (unit: mmol/mol) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  HbA1c.
Blood samples (unit: IU/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  FSH; LH.
Blood samples (unit: µg/L). | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  IGF-1.
Blood samples (unit: pmol/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  ACTH.
Blood samples (unit: 10E-3IU/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  Prolactin; TSH.
Blood samples (unit: nmol/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  SHBG; testosterone; T4; estradiol.
Blood samples (unit: mg/L) | Baseline and 16 weeks
  Standardised fasting morning blood samples will be drawn after the patient has been resting in a sitting position for 15 minutes.
  C-reactive protein (CRP).
Diurnal urine samples | Baseline and 16 weeks
  24 hours urine sampling are stored at -80C until analysis. Cortisol metabolites will be measured in nmol/24h.
Hair samples | Baseline and 16 weeks
  Two hair samples are collected. Each sample is a section of hair strands approximately 3 mm in diameter and cut as close as possible to the scalp with a scissor. The hair samples are collected from the posterior vertex area. The cut end of the hair strands is marked. The samples are stored in a dry and cool place for later analysis of hair cortisol levels.
Saliva samples | Baseline and 16 weeks
  Fasting saliva samples are collected to measure salivary cortisol.
Continous glucose monitoring (CGM) | Baseline and 16 weeks, duration: 7 days
  Patients will wear a Dexcom G6 sensor to measure glucose levels.
Muscle biopsies | Baseline and 16 weeks
  Patients attending Aarhus University Hospital will be requested to provide muscle and fat biopsies.
  During sterile conditions and local anaesthesia, muscle biopsies (≈ 500 mg) are obtained from the vastus lateralis of the quadriceps femoris muscle 10-15 cm proximal to the patella using a Bergström biopsy needle.
Fat biopsies | Baseline and 16 weeks
  Patients attending Aarhus University Hospital will be requested to provide muscle and fat biopsies.
  Adipose tissue biopsies (≈ 20 ml) are obtained by liposuction from the abdominal subcutaneous fat depots during local anaesthesia.
Physical examination - Height | Baseline and 16 weeks
  Height is measured in cm.
Physical examination - Weight | Baseline and 16 weeks
  Weight is measured in kg.
Physical examination - waist and hip circumference. | Baseline and 16 weeks
  Waist and hip circumference are measured in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S Andersen, Principal Investigator — Odense University Hospital
Locations (3):
- Denmark (3):
  - Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus
  - Department of Nephrology and Endocrinology, Rigshospitalet, Copenhagen
  - Department of Endocrinology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
Deidentified participant data will be made available after completion of the study and publication of the main results, upon reasonable request. Data sharing will comply with GDPR and national data protection regulations.

REFERENCES:
- [Derived] Dreyer AF, Hansen SB, Borresen SW, Al-Jorani H, Bislev LS, Boesen VB, Christensen LL, Glintborg D, Jensen RC, Jorgensen NT, Klose MC, Lund ML, Frederiksen JSS, Tei R, Feldt-Rasmussen U, Jorgensen JOL, Andersen MS. Hydrocortisone replacement therapy in patients with glucocorticoid withdrawal syndrome after cessation of glucocorticoid treatment: REPLACE, a multicentre, randomised, double-blinded, placebo-controlled, 16-week study protocol. BMJ Open. 2026 Feb 4;16(2):e111334. doi: 10.1136/bmjopen-2025-111334. PMID 41638742